CLINICAL TRIAL: NCT03522337
Title: Effectiveness of Visual Pedagogy-assisted Tooth-brushing Training Among Preschoolers With Special Needs for Oral Health Promotion
Brief Title: Oral Health Promotion Among Preschool Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Gloria Hai-Ming Wong, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCCC2016to2018; HKUCTR-2015 (Registry Identifier: HKU Clinical Trials Registry (HKUCTR))
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Intellectual Disability; Cerebral Palsy; Developmental Disorders; Developmental Delay; Autistic Spectrum Disorders; Down Syndrome; Epilepsy; Developmental Disability; Learning Disorders
Keywords: preschool children; special needs; tooth brushing; social story; visual pedagogy
MeSH Terms: conditions — Intellectual Disability; Cerebral Palsy; Developmental Disabilities; Learning Disabilities; Autism Spectrum Disorder; Down Syndrome; Epilepsy

STUDY DESIGN:
Intervention Model Description: This study is designed as a 24-month randomised, controlled, blind, parallel clinical trial conducted in Special Child Care Centres, aiming to promote oral health among preschool children with special needs.
Who Masked: Participant, Outcomes Assessor
Masking Description: The randomised sequence will be generated by an investigator who does not participate in the outreach service. The allocation sequence will be sealed in an envelope, and opened at the Special Child Care Centres by an assistant. The assistant will be responsible for delivering the materials to children and their parents.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The main intervention is conventional leaflets. Tooth-brushing training (toothbrushes and toothpastes provided) and oral health instruction are reinforced by leaflets.
  Interventions: Other: Conventional leaflets
- Test group (Experimental): The main intervention is visual pedagogy (social stories). Tooth-brushing training (toothbrushes and toothpastes provided) and oral health instruction are reinforced by social stories.
  Interventions: Other: Visual pedagogy (social stories)

INTERVENTIONS:
Other: Visual pedagogy (social stories) — Oral health instruction, tooth-brushing training (toothbrushes and fluoridated toothpastes provided)
  Other Names: Behavioral
  Arms: Test group
Other: Conventional leaflets — Oral health instruction, tooth-brushing training (toothbrushes and fluoridated toothpastes provided)
  Other Names: Behavioral
  Arms: Control group

SUMMARY:
Establishing good oral health-related habit is challenging among younger children, especially for preschool children with special needs, as they have physical, mental, sensory, behavioural, emotional, and chronic medical conditions that requires health care beyond the routines. Existing evidences showed that children with special needs have poorer oral health status and more challenging behaviours than their counterparts in main stream schools. Visual pedagogy, such as social stories, have been applied to teach a variety of skills or behaviours to individuals with special needs. They are short stories demonstrating the target skill or behaviour, and then the readers are expected to perform the target skill or behaviour following the demonstrations. Giving the evidence that children with special needs can understand complex situations and learn new practices by using those stories, we expect to apply a package of structured social stories to modify oral health-related behaviours (tooth brushing, healthy eating, dental visit), and thereby, improve oral health status among preschool children with special needs. Establishment of good oral-health related behaviours in early childhood will benefits children in their future life. Additionally, visual pedagogy-assisted oral health education is relatively easy and safe to implement. If proven effective, social story-based preventive care can be recommended to special children globally.

DETAILED DESCRIPTION:
Early childhood caries (ECC) is reported to be the most prevalent childhood disease. It is a chronic, infectious dental disease affecting children aged between birth and 71 months. Untreated ECC can lead to toothache, swelling, abscess, immature loss of primary teeth, and thereby, significant impacts on children's physical and emotional status. Nowadays, ECC has been recognised as a serious public health problem in developing as well as developed countries. Although ECC has a complex aetiology, existing evidence reveals that tooth brushing, appropriate eating habits, and regular dental check-ups are effective in preventing the development of ECC.

In this study, oral health education will be reinforced by a series of visual education materials (social stories or conventional leaflets), which covering the three topics in ECC prevention, namely "tooth brushing", "healthy diets", and "dental visit". Sample size calculation is performed by the program G* power 3.1.9.2. The primary outcome is the development of new dental caries over the 24-month study period. Clinical oral examinations will be performed according to the following criteria: i) Caries experiences were assessed by the International Caries Detection and Assessment System(ICDAS); ii) Oral hygiene status by Simplified oral hygiene index of Greene and Vermilion (OHI-S); iii) gingival health status by Modified Gingival Index of Lobene (MGI). Dental examination will be performed at Special Child Care Centres by a paediatric dentist with a disposable mouth-mirror attached to an LED light. Tell- Show-Do (TSD) technique will be used to improve children's cooperation level. Tooth-brushing performance will be assessed by two observers. After dental examination and tooth-brushing assessment, a standard hands-on tooth-brushing training will be provided immediately to each child and his/her parent. Oral health instruction will also be illustrated to the participants, reinforced by social stories (experiment group) or conventional leaflets (control group). Questionnaires regarding children's oral health related behaviours and family demographic information will be completed by parents, while children's developmental profile will be assessed by staff in Special Child Care Centres. Children' oral health status and expected behaviours (tooth brushing, healthy eating habits and dental-visit experience) will be assessed at 6-month, 12-month and 24-month intervals.

All the data will be analysed using IBM SPSS. Continuous valuables such as dmft, dmfs, S-OHI, MGI scores between the control and test groups will be analysed by two-sample t test, paired-t test, Mann-Whitney Test when appropriate. Chi-square statistics will be used to assess the differences in categorical variables between control group and test group, such as caries incidence, tooth-brushing frequencies, snacking frequencies, and dental-visit frequencies. McNemar's test will be used to analyse whether children's oral-health related behaviours will be changed before and after intervention. Regression analyses will be conducted to determine potential factors associated with children's oral health status or oral-health related behaviours in the model. The significance levels will be set to be P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Preschool-aged children in Special Child Care Centres or special schools in Hong Kong

Exclusion Criteria:

* With severe visually impaired, severe hearing impaired (cannot hear dentists' or parents' instruction); severe physical disabled (cannot hold a toothbrush); requiring emergent dental treatment; use of antibiotic within 3 months; dental prophylaxes in the last 6 months.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in carious tooth surfaces over course of the trial | The change from baseline to 24 months
  Assessed by the International Caries Detection and Assessment System(ICDAS)
Change in the prevalence of dental caries | The change from baseline to 24 months
  Measured by dmft index (decayed, missing due to caries, and filled primary teeth)

SECONDARY OUTCOMES:
Change in oral hygiene status | 6 months, 12 months, 24 months
  Assessed by simplified oral hygiene index (S-OHI)
Change in gingival status | 6 months, 12 months, 24 months
  Assessed by modified gingival index (MGI)
Change in children's tooth-brushing performance | 6 months, 12 months, 24 months
  Observed and assessed by investigators using the step-based assessment tool, and tooth-brushing duration will be recorded by a timer
Change in children's eating habits | 12 months, 24 months
  Questionnaires regarding children's oral health-related eating habits will be completed by parents
Change in children's dental-visit experience | 24 months
  Questionnaires regarding children's dental-visit experience will be completed by parents
The amount of toothpaste | Immediately after dentists demonstrating the appropriate amount of toothpaste for children younger than 6 years old
  The weight of toothpaste dispensed by parents and/or children during tooth-brushing training
Toothbrush wear | 6 months, 12 months, 24 months
  Assessed by toothbrush wear index (Rawls,1989)

CONTACTS AND LOCATIONS:
Overall Officials: Hai Ming Wong, PhD, Principal Investigator — Dental Faculty, The University of Hong Kong
Locations (1):
- Dental Faculty, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
After the relevant studies have been published, Statistical Analysis Plan and Clinical Study Report will be shared.
Supporting Information: SAP, CSR
Time Frame: Relevant date will be shared 6 months later after the summary data are published.
Access Criteria: E-mail

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03522337/SAP_000.pdf
  • Study Protocol (2015-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03522337/Prot_001.pdf